CLINICAL TRIAL: NCT00247182
Title: Stepped Care for Mandated College Students
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Brian Borsari, PI, National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NIAAABOR015518; NIH Grant R01 AA015518-01
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Alcohol Use
Keywords: Stepped Care; Brief Motivational Intervention; Minimal Intervention; Treatment response; College Students
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Step 1 (Other): Minimal Intervention
  Interventions: Behavioral: Step 1: Minimal Intervention; Behavioral: Step 2: Brief Motivational Intervention
- Step 2-A (Active Comparator): Brief motivational intervention (BMI)
  Interventions: Behavioral: Step 2: Brief Motivational Intervention
- Step 2-B (Active Comparator): Assessment-only control
  Interventions: Behavioral: Alcohol Assessment

INTERVENTIONS:
Behavioral: Step 1: Minimal Intervention — All participants will receive Step 1, a 15-minute minimal intervention including a discussion of the referral incident and the provision of a booklet containing advice to reduce drinking. Participants will be assessed six weeks later. All students will complete 3, 6, and 9 month follow-up assessments
  Arms: Step 1
Behavioral: Step 2: Brief Motivational Intervention — Participants continuing to exhibit risky alcohol use will receive Step 2, randomization to: (a) a 60-90 minute brief motivational intervention (BMI) or (b) an assessment-only control. All students will complete 3, 6, and 9 month follow-up assessments.
  Arms: Step 1; Step 2-A
Behavioral: Alcohol Assessment — Participants continuing to exhibit risky alcohol use will receive Step 2, randomization to: (a) a 60-90 minute brief motivational intervention (BMI) or (b) an assessment-only control. All students will complete 3, 6, and 9 month follow-up assessments.
  Arms: Step 2-B

SUMMARY:
This project provides stepped care to college students mandated for alcohol-related offenses. Students are first provided with a minimal intervention, a 15-minute discussion of their alcohol use. Students who continue to drink in a risky manner are provided with a more intensive, hour-long brief motivational interview. By providing more intensive treatment to the students who exhibit risky drinking, we hope to maximize the efficiency of campus alcohol programs.

DETAILED DESCRIPTION:
Colleges and universities have seen a large increase in the number of students referred to the administration for the violation of alcohol policies. However, research indicates that the majority of mandated students may not require extensive treatment. Stepped care assigns individuals to different levels of care according to their response to treatment. Encouraging research indicates that minimal interventions and BMIs may reduce heavy drinking in mandated college students. Thus, implementing stepped care using these interventions could maximize treatment efficiency and reduce the demands on campus alcohol programs.

Participants will be students mandated to attend an alcohol program at a northeastern private university. All participants will receive Step 1, a 15-minute minimal intervention including a discussion of the referral incident and the provision of a booklet containing advice to reduce drinking. Participants will be assessed six weeks later, and those continuing to exhibit risky alcohol use will receive Step 2, randomization to: (a) a 60-90 minute brief motivational intervention (BMI) or (b) an assessment-only control. All students will complete 3, 6, and 9 month follow-up assessments. The three groups will be compared on two outcome measures: frequency of binge drinking episodes and alcohol-related problems in the past 30 days. Predictors of treatment response (readiness to change, alcohol expectancies, age of first drink, sensation seeking, descriptive norms, and reaction to the referral) will also be evaluated for both steps of the intervention. Research findings will assist college alcohol programs in determining the most effective and efficient allocation of their limited resources in treating mandated students. The long-term objectives of this research are to inform preventive intervention research about the utility and cost-effectiveness of stepped-care approaches and to identify individual and situational factors that qualify these effects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female students 18 years of age or older.
* Participants will have signed a witnessed informed consent.
* Participants will have been referred for an alcohol-related offense

Exclusion Criteria:

* Participants who meet current DSM-IV criteria for substance use disorder
* Participants who are currently in treatment for substance use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2006-10; Primary Completion 2010-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | 3, 6, and 9 months
Alcohol-related consequences | 3, 6, and 9 months

SECONDARY OUTCOMES:
Predictors of response to treatment | 3, 6, and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian E. Borsari, PhD, Principal Investigator — Brown University
Locations (1):
- Roger Williams University, Bristol, Rhode Island, United States

REFERENCES:
- [Background] Borsari B, O'Leary Tevyaw T, Barnett NP, Kahler CW, Monti PM. Stepped care for mandated college students: a pilot study. Am J Addict. 2007 Mar-Apr;16(2):131-7. doi: 10.1080/10550490601184498. PMID 17453615
- [Background] Borsari B, Murphy JG, Barnett NP. Predictors of alcohol use during the first year of college: implications for prevention. Addict Behav. 2007 Oct;32(10):2062-86. doi: 10.1016/j.addbeh.2007.01.017. Epub 2007 Jan 23. PMID 17321059
- [Background] Borsari B, Muellerleile P. Collateral reports in the college setting: a meta-analytic integration. Alcohol Clin Exp Res. 2009 May;33(5):826-38. doi: 10.1111/j.1530-0277.2009.00902.x. Epub 2009 Mar 6. PMID 19298324
- [Result] Hustad JT, Eaton Short E, Borsari B, Barnett NP, O'Leary Tevyaw T, Kahler CW. College alcohol citations result in modest reductions in student drinking. J Subst Abuse Treat. 2011 Apr;40(3):281-6. doi: 10.1016/j.jsat.2010.11.005. Epub 2010 Dec 28. PMID 21193284
- [Result] Barthelmes CK, Borsari B, Hustad JT, Barnett NP. Hostility in mandated students: exploratory analysis and implications for treatment. J Subst Abuse Treat. 2010 Apr;38(3):284-91. doi: 10.1016/j.jsat.2010.01.004. Epub 2010 Feb 8. PMID 20116962
- [Result] Barnett NP, Borsari B, Hustad JT, Tevyaw TO, Colby SM, Kahler CW, Monti PM. Profiles of college students mandated to alcohol intervention. J Stud Alcohol Drugs. 2008 Sep;69(5):684-94. doi: 10.15288/jsad.2008.69.684. PMID 18781243
- [Result] Kahler CW, Hustad J, Barnett NP, Strong DR, Borsari B. Validation of the 30-day version of the Brief Young Adult Alcohol Consequences Questionnaire for use in longitudinal studies. J Stud Alcohol Drugs. 2008 Jul;69(4):611-5. doi: 10.15288/jsad.2008.69.611. PMID 18612578
- [Result] Borsari B, Boyle KE, Hustad JT, Barnett NP, O'Leary Tevyaw T, Kahler CW. Drinking before drinking: pregaming and drinking games in mandated students. Addict Behav. 2007 Nov;32(11):2694-705. doi: 10.1016/j.addbeh.2007.05.003. Epub 2007 May 17. PMID 17574344
- [Result] Borsari B, Hustad JT, Mastroleo NR, Tevyaw TO, Barnett NP, Kahler CW, Short EE, Monti PM. Addressing alcohol use and problems in mandated college students: a randomized clinical trial using stepped care. J Consult Clin Psychol. 2012 Dec;80(6):1062-74. doi: 10.1037/a0029902. Epub 2012 Aug 27. PMID 22924334
- [Result] Borsari B, Short EE, Mastroleo NR, Hustad JT, Tevyaw TO, Barnett NP, Kahler CW, Monti PM. Phone-delivered brief motivational interventions for mandated college students delivered during the summer months. J Subst Abuse Treat. 2014 May-Jun;46(5):592-6. doi: 10.1016/j.jsat.2014.01.001. Epub 2014 Jan 13. PMID 24512944
- [Result] Teeters JB, Borsari B, Martens MP, Murphy JG. Brief Motivational Interventions Are Associated With Reductions in Alcohol-Impaired Driving Among College Drinkers. J Stud Alcohol Drugs. 2015 Sep;76(5):700-9. doi: 10.15288/jsad.2015.76.700. PMID 26402350
- [Result] Yurasek AM, Borsari B, Magill M, Mastroleo NR, Hustad JT, Tevyaw TO, Barnett NP, Kahler CW, Monti PM. Descriptive norms and expectancies as mediators of a brief motivational intervention for mandated college students receiving stepped care for alcohol use. Psychol Addict Behav. 2015 Dec;29(4):1003-11. doi: 10.1037/adb0000092. Epub 2015 Jun 22. PMID 26098125
- [Result] Borsari B, Magill M, Mastroleo NR, Hustad JT, Tevyaw TO, Barnett NP, Kahler CW, Eaton E, Monti PM. Mandated college students' response to sequentially administered alcohol interventions in a randomized clinical trial using stepped care. J Consult Clin Psychol. 2016 Feb;84(2):103-12. doi: 10.1037/a0039800. Epub 2015 Oct 12. PMID 26460571
- [Derived] Fernandez AC, Yurasek AM, Merrill JE, Miller MB, Zamboanga BL, Carey KB, Borsari B. Do brief motivational interventions reduce drinking game frequency in mandated students? An analysis of data from two randomized controlled trials. Psychol Addict Behav. 2017 Feb;31(1):36-45. doi: 10.1037/adb0000239. Epub 2016 Dec 12. PMID 27936818
- See also: Related Info — http://research.brown.edu/research/profile.php?id=1128622883